CLINICAL TRIAL: NCT00435539
Title: A Randomized, Sham-Injection Controlled, Double-Masked, Ascending-Dose, Dose-Range-Finding Trial of Microplasmin Intravitreal Injection for Non-Surgical Posterior Vitreous Detachment (PVD) Induction for Treatment of Vitreomacular Traction (VMT).
Brief Title: A Study to Compare Multiple Doses Intravitreal Microplasmin for Treatment of Patients With Vitreomacular Traction (MIVI-IIt)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-MV-004; MIVI-IIT
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Results first posted 2013-09-13 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-04

CONDITIONS: Vitreomacular Traction
Keywords: Vitreomacular Traction; Maculopathy; VMT; PVD
MeSH Terms: conditions — Macular Degeneration | interventions — microplasmin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ocriplasmin 75µg single injection (Experimental): Ocriplasmin 75µg single injection versus sham injection
  Interventions: Drug: ocriplasmin
- ocriplasmin 125µg single injection (Experimental): Ocriplasmin 125µg single injection versus sham injection
  Interventions: Drug: ocriplasmin
- ocriplasmin 175µg single injection (Experimental): Ocriplasmin 175µg single injection versus sham injection
  Interventions: Drug: ocriplasmin
- ocriplasmin 125µg multiple injections (Experimental): Ocriplasmin 125µg multiple injections. Subjects who did not achieve resolution of VMT by the day 28 visit (i.e. non-responders) were given an open-label injection of ocriplasmin 125µg. Subjects who still did not achieve resolution of VMT by the day 56 visit were given a second open-label injection of ocriplasmin 125µg.
  Interventions: Drug: ocriplasmin
- sham injection (Sham Comparator): sham injection
  Interventions: Drug: Sham Comparator

INTERVENTIONS:
Drug: ocriplasmin — Intravitreal injection of ocriplasmin solution containing 75µg of ocriplasmin.
  Other Names: microplasmin
  Arms: ocriplasmin 125µg single injection; ocriplasmin 175µg single injection; ocriplasmin 75µg single injection
Drug: ocriplasmin — Intravitreal injection of ocriplasmin solution containing 125µg of ocriplasmin with up to 2 additional (open label) 125µg ocriplasmin injection at 1 month interval.
  Other Names: microplasmin
  Arms: ocriplasmin 125µg multiple injections
Drug: Sham Comparator — Intravitreal sham injection
  Other Names: microplasmin
  Arms: sham injection

SUMMARY:
A multicenter study to compare multiple doses of intravitreal microplasmin for non-surgical PVD induction for treatment of patients with vitreomacular traction.

ELIGIBILITY:
Inclusion Criteria:

* Patients >_ 18 years of age with vitreomacular traction

Exclusion Criteria:

* PVD present at baseline
* Certain vitreoretinal conditions including proliferative disease, rhegmatogenous retinal detachment, and proliferative vitreoretinopathy (PVR)
* Vitreous hemorrhage
* Patients who have had a vitrectomy in the study eye at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (3):
  - ZNA OCMW Antwerpen, Antwerp
  - University Hospital of Ghent, Ghent
  - Universitaire Ziekenhuizen K.U.Leuven, Leuven
- Augenklinik der Universitat Munchen, München, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was enrolled on 2 March 2007 and the last patient completed the last visit on 8 January 2009. All patients were selected in medical clinics
Pre-assignment Details: All subjects in all cohorts had a similar follow-up schedule to the day 28 post-injection visit. After day 28, non-responders in cohort 4 received up to 2 repeated injections and thus had a different study follow-up schedule than all other subjects.
Groups:
- Ocriplasmin 125µg Multiple Injections: ocriplasmin 125µg multiple injections. Subjects who did not achieve resolution of VMT by the day 28 visit (i.e. non-responders) were given an open-label injection of ocriplasmin 125 μg. Subjects who still did not achieve resolution of VMT by the day 56 visit were given a second open-label injection of ocriplasmin 125 μg.
Period: Overall Study
Arm/Group | Ocriplasmin 75µg Single Injection | Ocriplasmin 125µg Single Injection | Ocriplasmin 175µg Single Injection | Ocriplasmin 125µg Multiple Injections | Sham Injection
Started | 12 | 13 | 11 | 12 | 12
Completed | 12 | 13 | 11 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ocriplasmin 125µg Multiple Injections: ocriplasmin 125µg multiple injections Subjects who did not achieve resolution of VMT by the day 28 visit (i.e. non-responders) were given an open-label injection of ocriplasmin 125 μg. Subjects who still did not achieve resolution of VMT by the day 56 visit were given a second open-label injection of ocriplasmin 125 μg.
- Total: Total of all reporting groups
Arm/Group | Ocriplasmin 75µg Single Injection | Ocriplasmin 125µg Single Injection | Ocriplasmin 175µg Single Injection | Ocriplasmin 125µg Multiple Injections | Sham Injection | Total
Number analyzed (Participants) | 12 | 13 | 11 | 12 | 12 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.58 (5.57) | 74.67 (5.78) | 66.11 (9.08) | 70.61 (6.67) | 70.28 (8.58) | 69.79 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 4 | 7 | 6 | 33
  Male | 4 | 5 | 7 | 5 | 6 | 27

OUTCOME MEASURES:

1. Secondary Outcome: Resolution of Vitreomacular Traction (Investigator's Assessment)
Description: Resolution of VMT was evaluated by the investigator using optical coherence tomography (OCT).Resolution of VMT was defined as a change from baseline status of Yes to post-injection status of No and was evaluated by the investigator using OCT. Subjects undergoing vitrectomy had their last observation prior to vitrectomy carried forward.
Time Frame: Day 28
Population: Intention to Treat (ITT)
Measure: Number; unit: Percentage of participants
Groups:
- Ocriplasmin 125µg Pooled: Pooled data for ocriplasmin 125µg and ocriplasmin 125µg multiple injections versus sham injection
Arm/Group | Ocriplasmin 75µg Single Injection | Ocriplasmin 175µg Single Injection | Ocriplasmin 125µg Pooled | Sham Injection
Number analyzed (Participants) | 12 | 11 | 25 | 12
Percentage of participants | 25 | 27.3 | 11 | 8.3
Statistical Analysis 1: Comparison: Ocriplasmin 75µg Single Injection vs Sham Injection; Test type: Superiority or Other; p = 0.4783, Fisher Exact
Statistical Analysis 2: Comparison: Ocriplasmin 175µg Single Injection vs Sham Injection; Test type: Superiority or Other; p = 0.0932, Fisher Exact
Statistical Analysis 3: Comparison: Ocriplasmin 125µg Pooled vs Sham Injection; Test type: Superiority or Other; p = 0.0721, Fisher Exact

2. Primary Outcome: Proportion of Subjects With Total PVD at the First Day 14 Post-injection Visit (Vitreous Detachment to the Equator) as Determined by Masked Central Reading Center (CRC) Evaluation of B-scan Imaging.
Time Frame: Day 14
Population: Intention to Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Ocriplasmin 75µg Single Injection | Ocriplasmin 175µg Single Injection | Ocriplasmin 125µg Pooled | Sham Injection
Number analyzed (Participants) | 11 | 11 | 22 | 11
percentage of participants | 18.2 | 18.2 | 13.6 | 0
Statistical Analysis 1: Comparison: Ocriplasmin 75µg Single Injection vs Sham Injection; Test type: Superiority or Other; p = 0.4762, Fisher Exact
Statistical Analysis 2: Comparison: Ocriplasmin 175µg Single Injection vs Sham Injection; Test type: Superiority or Other; p = 0.4762, Fisher Exact
Statistical Analysis 3: Comparison: Ocriplasmin 125µg Pooled vs Sham Injection; Test type: Superiority or Other; p = 0.5343, Fisher Exact

ADVERSE EVENTS:
Time Frame: AEs/SAEs were collected from injection day up to 6 months after injection
Groups:
- Ocriplasmin 75µg: Ocriplasmin 75µg single injection versus sham injection
- Ocriplasmin 125µg Multiple Injection: Ocriplasmin 125µg multiple injection versus sham injection
Arm/Group | Ocriplasmin 75µg | Ocriplasmin 125µg Single Injection | Ocriplasmin 175µg Single Injection | Ocriplasmin 125µg Multiple Injection | Sham Injection
Serious Adverse Events (participants affected / at risk) | 3/12 | 2/13 | 3/11 | 4/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 10/13 | 10/11 | 11/12 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 75µg (N=12) | Ocriplasmin 125µg Single Injection (N=13) | Ocriplasmin 175µg Single Injection (N=11) | Ocriplasmin 125µg Multiple Injection (N=12) | Sham Injection (N=12)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Silent Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocriplasmin 75µg (N=12) | Ocriplasmin 125µg Single Injection (N=13) | Ocriplasmin 175µg Single Injection (N=11) | Ocriplasmin 125µg Multiple Injection (N=12) | Sham Injection (N=12)
Vitreous floaters (Eye disorders) | 4 (4) | 3 (3) | 4 (4) | 7 (9) | 0 (0)
Vitritis (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Conjuctival hyperaemia (Eye disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Anterior chamber flare (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (3)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Macular pseudohole (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anterior chamber cell (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macular scar (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Maculopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meibomianitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic nerve cupping (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papilloedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous opacities (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ostheoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Endocrine disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less